CLINICAL TRIAL: NCT07337005
Title: CompREhensive Diagnostic Assessment of Coronary Endothelial Function Impairment and Vasospasm With CoNtinuous ThErmodilution in Patients With Suspected Coronary Microvascular and Vasomotor Dysfunction
Acronym: REDEFINE-CMD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRAS 356198
Record Dates: First submitted 2025-12-18; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Coronary Microvascular Dysfunction (CMD); Vasospasm, Coronary
MeSH Terms: conditions — Coronary Vasospasm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Invasive Coronary function Assessment arm (Experimental): Invasive coronary endothelial function and vasospasm assessment
  Interventions: Procedure: Invasive coronary physiological measurements

INTERVENTIONS:
Procedure: Invasive coronary physiological measurements — Invasive assessment of changes in coronary blood flow, resistance, and distal pressure in response to acetylcholine infusion. These will be measured during a clinical indicated invasive coronary angiogram procedure and physiological studies using a standard coronary pressure wire and a dedicated infusion catheter.

SUMMARY:
The goal of this observational study is to learn more about the diagnosis of coronary endothelium function and coronary vasospasm using a dedicated invasive protocol in patients who has angina without obstruction in their main heart arteries. The main question it aims to answer is the feasibility, reproducibility, and safety of this invasive protocol:

Does this invasive protocol diagnose coronary endothelial dysfunction and vasospasm without issues?

Participants already having invasive coronary angiogram and physiological studies will undergo additional physiological measurements during the same procedure.

Participants will enrol in a symptoms and quality of life questionnaire using dedicated questionnaires and a mobile application to assess the burden of their symptoms before and after the invasive procedure and up to 12 months follow up.

A subset of participants will undergo a repeat set of these measurements to assess reproducibility of the invasive protocol.

A subset of the participants will also undergo a cardiac MRI to assess correlation with the invasive protocol measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptoms suggestive of angina.
2. Evidence of unobstructed coronary arteries on invasive or non-invasive coronary angiography (coronary stenosis <50% and /or FFR >0.80).
3. Above the age of 18.
4. The subject has been informed of the nature of the study, agrees to its provisions and has signed written informed consent.

Exclusion Criteria:

1. Pregnancy.
2. Contraindication to angiography and/or physiological assessment with adenosine or acetylcholine.
3. Previous coronary artery bypass graft (CABG).
4. Moderate to severe valvular heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcome | At baseline
  Proportion of patients in whom the full invasive protocol (baseline and post-stimulation measurements) is successfully completed without major technical issues or protocol deviations.

SECONDARY OUTCOMES:
Reproducibility outcome | At baseline
  Intra- and inter-operator variability of measurements quantified using intraclass correlation coefficients and Bland-Altman plots in a predefined reproducibility subset.
Safety outcome | At Baseline and up to 12 months
  Incidence of adverse events related to the procedure or medications.
Correlation between invasive and non-invasive measures of endothelial-dependent coronary microvascular dysfunction. | From baseline and up to 3 months
  Strength of correlation (unit of measure = correlation coefficient, r) between invasive indices of endothelial-dependent coronary microvascular function obtained during the study protocol (absolute coronary blood flow and absolute microvascular resistance measured by continuous thermodilution during intracoronary acetylcholine testing) and non-invasive measures of myocardial perfusion (myocardial perfusion reserve obtained from cardiac stress perfusion imaging). Diagnostic agreement for identifying endothelial-dependent microvascular dysfunction will also be assessed (unit of measure = area under ROC curve, sensitivity, and specificity), using the invasive assessment as the reference standard.
Correlation between invasive physiological indices of coronary microvascular function and symptom burden at baseline. | Baseline (at time of invasive coronary function testing).
  The strength of correlation (Pearson or Spearman correlation coefficient; unit of measure = correlation coefficient, r) between invasive physiological measurements of coronary microvascular function obtained during the study protocol (e.g., absolute coronary blood flow and absolute microvascular resistance derived by continuous thermodilution during acetylcholine testing) and patient-reported symptom burden assessed at baseline using validated questionnaires (Seattle Angina Questionnaire-7 [SAQ-7] and EQ-5D-5L scores).
Change in symptoms, quality of life, and need for further investigation or treatment during follow-up. | From baseline to 12 months follow-up
  Change from baseline to follow-up in patient-reported symptoms and quality of life (unit of measure = change in questionnaire score) as assessed using the SAQ-7 and EQ-5D-5L questionnaires, and the proportion of patients (%) requiring additional cardiac investigations or treatment changes during follow-up.

IPD SHARING:
Plan to Share IPD: Undecided